CLINICAL TRIAL: NCT00856440
Title: Safety and Efficacy of Routine Colonoscopy Preparations
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Korsten, Mark - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B4162C-1; 2380-06-031
Record Dates: First submitted 2009-03-02; First posted 2009-03-05 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Spinal Cord Injury
Keywords: SCI
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Golytely

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: SCI
  Interventions: Drug: Fleets Oral Sodium Phosphate Solution (OSPS); Drug: Colyte; Drug: Dual (OSPS & Colyte)
- 2: Able-bodied
  Interventions: Drug: Fleets Oral Sodium Phosphate Solution (OSPS); Drug: Colyte; Drug: Dual (OSPS & Colyte)

INTERVENTIONS:
Drug: Fleets Oral Sodium Phosphate Solution (OSPS) — Osmotic preparation for colonoscopy
  Other Names: Phospho Soda
Drug: Colyte — Lavage preparation for colonoscopy
  Other Names: Golytely
Drug: Dual (OSPS & Colyte) — Combined, two-day preparation utilizing both preparations

SUMMARY:
Periodic screening for colon cancer has become the standard of care in individuals over the age of 50. In this context, it is generally accepted that colonoscopy is the most sensitive modality for the detection of colon cancer and/or pre malignant colon pathology. As currently performed, however, colonoscopy requires that stool be eliminated from the colon before the examination. If stool remains in the colon, visualization of the bowel will be partially or completely impaired and limits the effectiveness of the screening. A number of methods are employed for purging the bowel of waste material but they generally involve either administration of a lavage (like a flush) solution (such as Colyte or Golytely) or of an osmotic laxative (such as sodium phosphate or magnesium citrate). Neither of these approaches is uniformly effective in all individuals and neither is without potential complications, especially on the kidneys. It is the intent of the proposed research to study the relative efficacy and safety of these preparations in both able-bodied individuals as well as people with spinal cord injury. To this end, we will randomize these groups to a lavage solution, a laxative or a combination of the two prior to a routine, clinically indicated colonoscopy. The quality of the preparation will be directly assessed during the colonoscopy and the effect of these preparations on kidney function will be determined. We suspect that when it comes to preparation for colonoscopy, one shoe does not fit all sizes. The proposed research should allow us to determine which form of preparation is least harmful while achieving optimal effectiveness.

DETAILED DESCRIPTION:
Colonoscopy is a routine evaluation for screening of colorectal cancer in people over 50 and for those at increased genetic risk. Despite the large number of individuals requiring such screening, there has been little randomized, controlled research to determine the relative renal safety of oral colon preparation solutions that are used to evacuate the bowel in patients with "normal" kidney function, the best frequency of laxative dosing (e.g. 1 day vs. 2 day), and the quality of the colon cleansing that results from these different approaches. Reports of acute renal failure, secondary to nephrocalcinosis, following the commonly used oral phosphosoda preparation are increasingly recognized. It is our belief that this project will yield clinically relevant information that would have immediate clinical application for all persons receiving a colonoscopy. Since preparation for screening colonoscopy involves vigorous purging of stool from individuals without GI complaints, it also represents an opportunity to study the prevalence of clostridium difficile (C. diff) in this population. This may reveal important information regarding the epidemiology of this increasingly virulent and common enteric pathogen. A pilot screening program for asymptomatic C. diff, a common nosocomial pathogen, may reveal findings of clinical importance for preventing spread of this infection, and allow use of presumptive treatment during periods of increased risk.

ELIGIBILITY:
Inclusion Criteria:

1. Patients already clinically indicated for colonoscopy examination

Exclusion Criteria:

1. Patients who are not a candidate for elective colonoscopy (i.e. those with recent myocardial infarction, terminal illness, etc.)
2. Patients who have a contraindication for Colyte (i.e. those with colonic obstruction, etc.)
3. Patients who have a contraindication for Fleet OSPS (i.e. those with poor renal function, class 2 or greater symptomatic heart failure, etc.)
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans, SCI and able-bodied
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2006-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Renal Function (GFR, creatinine clearance) | <30 days

SECONDARY OUTCOMES:
Quality of bowel preparation (Ottawa Score) | <30 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Korsten, MD, Principal Investigator — VA Medical Center, Bronx
Locations (1):
- VA Medical Center, Bronx, The Bronx, New York, United States